CLINICAL TRIAL: NCT01416922
Title: The oncoFISH Cervical Test for Detection of 3q26 Region Gain
Brief Title: oncoFISH Cervical Test for Detection of 3q26 Region Gain
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Ikonisys, Inc. (Industry)
Responsible Party: CEO, Ikonisys
Other Study IDs: IKON 0801; NCT01417039 (obsolete NCT alias)
Record Dates: First submitted 2011-08-12; First posted 2011-08-15 (Estimated); Last update posted 2011-08-15 (Estimated); Status verified 2011-08

CONDITIONS: Cervical Cancer; LSIL
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- LSIL: Women 21 years of age or older with an LSIL diagnosis

SUMMARY:
The purpose of this study is to evaluate the use of the oncoFISH cervical test system in the management of women who have received an LSIL Pap report to determine whether the test can predict which women will progress to more serious cervical disease and which women do not have to be monitored as closely.

ELIGIBILITY:
Inclusion Criteria:

* Women 21 years of age or greater with recent LSIL who are scheduled for colposcipal assessment.
* Women with previous or current STD or HIV may be included
* Women with previous LSIL history may be included.

Exclusion Criteria:

* pregnant women,
* women with vaginal intraepithelial lesions,
* women on a chemotherapeutic agent,
* women with previous or current cancer except for non-cervical squamous cell carcinoma

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients 21 years of age or greater with LSIL cytology diagnosis who are scheduled for a colposcical assessment.
Sampling Method: Probability Sample
Enrollment: 1100 (Estimated)
Dates: Start 2009-06; Study Completion 2011-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Michael W Kilpatrick, Ph.D., Study Director — Ikonisys, Inc.
Locations (1):
- Ikonisys, New Haven, Connecticut, United States